CLINICAL TRIAL: NCT07246577
Title: The VGR GCA Cohort
Brief Title: The VGR GCA Cohort: Ultrasound, Biopsy and Biomarkers - Novel Methods for Diagnosis, Monitoring and Prognosis in Giant Cell Arteritis.
Status: Not yet recruiting | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-02518-01
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Giant Cell Arteritis (GCA)
Keywords: Prospective Studies; Validation Study; Giant Cell Arteritis; Ultrasonography; Biomarkers; Temporal Arteries; Biopsy
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples including serum, plasma, whole blood, and tissue (temporal artery biopsy) will be collected.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GCA group: Individuals diagnosed with GCA
- Control group: Individuals not diagnosed with GCA

SUMMARY:
Giant cell arteritis (GCA) is the most common vasculitis in the elderly and is usually treated with long-term corticosteroid therapy. Many patients experience relapses and treatment-related side effects. Current diagnostic and monitoring methods provide limited prognostic information and cannot reliably distinguish active from inactive disease during relapse. This project addresses the clinical need for improved tools to identify patients at high risk of relapse and to develop more effective methods for disease monitoring.

The aim is to develop new tools that enable more personalized treatment of GCA. By combining vascular ultrasound with novel blood biomarkers, we seek to predict disease course and relapse risk. The specific objectives are:

* To identify ultrasound and blood biomarkers that can predict long-term disease control.
* To determine which ultrasound parameters and blood biomarkers can distinguish active from inactive disease during treatment.
* To evaluate whether extended vascular ultrasound protocols can improve diagnostic accuracy.

The ultimate goal is to establish safe, practical tools for improved diagnosis and follow-up in patients with GCA.

DETAILED DESCRIPTION:
Background Giant cell arteritis (GCA) is the most common form of vasculitis in older adults and is characterized by inflammation of medium- and large-sized arteries. The disease can cause serious complications such as vision loss, aortic aneurysm, and stroke. Treatment is mainly based on long-term glucocorticoid therapy. Despite this, 30-60% of patients experience disease relapse during treatment, and many develop steroid-related side effects. There are substantial knowledge gaps regarding optimal treatment stratification, reliable differentiation between active inflammation and chronic vascular remodeling, and the ideal extent of vascular ultrasound examination for diagnostic accuracy.

Overall Aim and Specific Objectives The overarching aim of this study is to determine which ultrasound parameters and novel blood biomarkers have prognostic, monitoring, and diagnostic value in GCA. The goal is to enable more individualized therapy and to reduce the risk of both over- and undertreatment.

Specific objectives are:

* To identify ultrasound parameters and biomarkers with prognostic value for long-term treatment response.
* To identify ultrasound parameters and biomarkers that distinguish active from inactive inflammation during treatment and at diagnosis.
* To evaluate whether an extended vascular ultrasound protocol improves diagnostic accuracy compared with the current European (EULAR) recommendations, and to assess whether ultrasound-detected neovascularization corresponds to histological neovascularization in temporal artery biopsy specimens.

Current Research Context Diagnostic advances in GCA have recently been driven by imaging techniques, particularly ultrasound. The European Alliance of Associations for Rheumatology (EULAR) currently recommends ultrasound assessment of the temporal and axillary arteries in suspected GCA. Quantitative parameters such as intima-media thickness (IMT) and scoring systems (e.g., Halo count and the OMERACT GCA Ultrasonography Score, OGUS) are used to assess vascular wall inflammation. However, these methods primarily evaluate cranial arteries and the axillary arteries. Studies using PET-CT have shown that extracranial vascular involvement is common and associated with a higher relapse risk and longer treatment duration. We have previously developed an extended ultrasound protocol that includes a broader set of extracranial arteries. In a retrospective study, we demonstrated that this extended protocol improves diagnostic accuracy compared to the EULAR-recommended approach.

Distinguishing active inflammation from chronic vascular alterations remains difficult. IMT may remain thickened even after resolution of inflammation. Neovascularization, detectable using modern low-flow ultrasound software, reflects microcirculation and angiogenesis in the vessel wall. Recent studies have demonstrated that neovascularization can be visualized in smaller temporal arteries in patients with active GCA, and that its presence correlates with more extensive disease. Neovascularization thus appears to represent a morphological marker of active inflammation. These previous data together with findings from Takayasu arteritis suggest that ultrasound-detected neovascularization could complement IMT as a sensitive indicator of disease activity. Based on these insights, we aim to integrate both IMT and neovascularization into a composite ultrasound score with potential prognostic and monitoring value.

Currently, disease activity in GCA is primarily assessed using CRP and ESR, which have limited sensitivity and specificity, especially in patients treated with IL-6 inhibitors. Novel biomarkers directly linked to vascular wall inflammation and destruction have been identified in experimental models. Interleukin-9 (IL-9) has been shown to promote inflammation and vascular injury in GCA models, while IL-9 blockade reduces disease severity. Angiopoietin-2 is involved in angiogenesis, and matrix metalloproteinase-3 (MMP-3) contributes to vascular wall degradation. These biomarkers are promising but have not yet been evaluated in clinical GCA cohorts.

A total of 100 individuals with GCA are required for the primary outcome, assuming an alpha level of 0.05, a power of 0.90, and an estimated dropout rate of 25%. Based on an estimated GCA prevalence of 30% among referred patients, approximately 340 ultrasound examinations will be needed to achieve the target sample size.

In summary, diagnostic imaging of GCA has advanced considerably through ultrasound, yet the prognostic and monitoring applications of this technique remain largely unexplored, particularly in combination with novel vascular biomarkers. This study will integrate advanced vascular ultrasound with biomarker analyses to improve diagnostic precision, disease monitoring, and individualized treatment strategies in GCA.

ELIGIBILITY:
Inclusion Criteria

* Individuals referred for evaluation due to suspected giant cell arteritis (GCA).
* Ability to provide written informed consent.

Exclusion Criteria

* Previous diagnosis of GCA.
* Previous temporal artery biopsy performed as part of prior GCA evaluation.
* Treatment with high-dose corticosteroids (>7.5 mg/day) for more than two weeks before initiation of the diagnostic work-up.
* Inability to provide informed consent.
* Inability to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A new cohort will be recruited. Individuals presenting with suspected GCA at Sahlgrenska University Hospital in Gothenburg, Sweden, or at Skaraborg Hospital Skövde, Sweden, will be invited to participate in the study. Diagnostic ultrasound examinations and follow-up assessments will be conducted at Sahlgrenska University Hospital in Gothenburg. After study enrollment, participants diagnosed with GCA will be followed for 12 months, with scheduled visits at 1, 6, and 12 months after initiation of treatment. If clinical relapse of GCA is suspected outside of the scheduled visits, an additional examination will be performed. Participants who are not diagnosed with GCA will be followed up by telephone after 6 months to confirm diagnostic status.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Sustained remission | 12 months
  Defined as achievement of a daily glucocorticoid dose of ≤5 mg after 12 months of standardized treatment according to the treatment protocol recommended by the Swedish Society for Rheumatology.
  Primary Objective:
  To determine which ultrasound parameters and novel biomarkers, individually and as a composite measure (intima-media thickness [IMT] + morphological neovascularization), have prognostic value for remission and relapse in patients with giant cell arteritis (GCA).
  Primary Hypotheses:
  1a. The composite measure (IMT + morphological neovascularization) predicts remission at 12 months more accurately than each individual parameter or previously established ultrasound metrics.
  1b. Clinically applicable threshold values exist for the composite measure and for selected biomarkers that distinguish patients achieving remission from those who do not.

SECONDARY OUTCOMES:
Relapse | Up to 12 months
  Defined as recurrence of symptoms attributable to GCA (after exclusion of alternative causes) and/or erythrocyte sedimentation rate (ESR) ≥30 mm/h and C-reactive protein (CRP) ≥10 mg/L, with improvement of symptoms and/or ESR or CRP following escalation of anti-inflammatory therapy.
  Secondary Objectives (1):
  To identify ultrasound parameters and biomarkers that best differentiate active from inactive vascular inflammation during ongoing GCA treatment in patients with suspected relapse.
  Secondary Hypotheses (1):
  1a. Changes in neovascularization, alone or combined with IMT, correlate more strongly with clinically defined relapse than changes in IMT alone.
  1b. The combination of ultrasound parameters and biomarkers provides higher diagnostic accuracy (AUC) for distinguishing active from inactive disease during treatment follow-up than current standard measures.
Final Diagnosis of GCA | 6 months
  Final diagnosis is based on clinical and imaging criteria in accordance with the 2022 American College of Rheumatology/European Alliance of Associations for Rheumatology (ACR/EULAR) classification criteria for GCA. Diagnosis will be re-evaluated after 6 months.
  Secondary Objectives (2):
  To evaluate whether an extended vascular ultrasound protocol (beyond temporal and axillary arteries) improves diagnostic accuracy compared to current EULAR recommendations, and whether ultrasound-detected neovascularization corresponds to histological neovascularization in temporal artery biopsy specimens.
  Secondary Hypotheses (2):
  2a. The extended ultrasound protocol increases sensitivity for GCA diagnosis without reducing specificity compared with the standard protocol.
  2b. Ultrasound-detected neovascularization corresponds with histological findings of angiogenesis in temporal artery biopsy samples (reference test).

CONTACTS AND LOCATIONS:
Locations (1):
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that underlie the results reported in publications arising from this study will be shared, after de-identification. This includes clinical, imaging, and biomarker data directly supporting the primary and secondary outcomes.
Supporting Information: Study Protocol
Time Frame: IPD and supporting documents will be made available starting 6 months after publication of the primary endpoint results and will remain accessible for 2 years thereafter.
Access Criteria: De-identified individual participant data and supporting materials will be available to qualified researchers upon reasonable request for purposes of meta-analysis or secondary research consistent with the study objectives. Requests will be reviewed by the principal investigator, and data will be shared through a secure data transfer process following approval.